CLINICAL TRIAL: NCT07384897
Title: Immune Cells Role in Lung Cancer and Their Use in Anticancer Immunotherapies and Inflammatory Lung Disease
Acronym: IMMUNOPUMON2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IMMUNOPOUMON2
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer (Diagnosis); Sarcoidosis; Chronic Obstructive Pulmonary Disease; Immunotherapy Resistance; Immune Dysregulation
Keywords: lung cancer; Non-Small Cell Lung Cancer; Sarcoidosis; Chronic Obstructive Pulmonary Disease; COPD; Immune Cells; Tumor Microenvironment; Immune Dysregulation; Immunotherapy; Immunotherapy Resistance; Immune Profiling; Myeloid Cells; Neutrophils; Dendritic Cells; Inflammation; Chronic Inflammation; Immune suppression; Emergency myelopoiesis
MeSH Terms: conditions — Lung Neoplasms; Disease; Sarcoidosis; Pulmonary Disease, Chronic Obstructive; Carcinoma, Non-Small-Cell Lung; Inflammation

STUDY DESIGN:
Intervention Model Description: This is a translational, non-interventional study evaluating immune cell populations in patients with lung cancer, sarcoidosis, and COPD. Participants receive only standard clinical care; no experimental treatments are given. Biological samples (primarily blood and when available, tumor, bone morrow samples collected for clinical reasons) and associated clinical data are analyzed to investigate immune mechanisms related to tumor progression, chronic lung inflammation, and response or resistance to therapy. The study is exploratory and comparative across diseases. All treatment decisions are made independently by the treating physicians and are not influenced by study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Patients with precancerous lung lesions (Other): Patients with precancerous lung lesions under clinical monitoring
  Interventions: Other: Peripheral Blood Collection for Immune Profiling
- Lung cancer (Active Comparator): Patients with a diagnosis of lung cancer (all stages)
  Interventions: Other: Peripheral Blood Collection for Immune Profiling
- Sarcoidosis and COPD (Other): Patients with chronic inflammatory lung diseases
  Interventions: Other: Peripheral Blood Collection for Immune Profiling
- Control group (Other): Control group of volunteers without known lung disease
  Interventions: Other: Peripheral Blood Collection for Immune Profiling
- chronic granulomatous disease (Other): Children and adolescents weighing ≥10 kg with chronic granulomatous disease
  Interventions: Other: Peripheral Blood Collection for Immune Profiling
- Adults undergoing orthopedic surgery following hip or femur fracture (Other): Bone Marrow of Adults undergoing orthopedic surgery following hip or femur fracture
  Interventions: Other: Peripheral Blood Collection for Immune Profiling

INTERVENTIONS:
Other: Peripheral Blood Collection for Immune Profiling — Participants provide biological samples for immune profiling and translational research. Samples include peripheral blood and, when available from routine clinical care, additional specimens such as tumor tissue or rlymph node, bone marrow. No experimental treatments are given. Collected samples are analyzed to characterize immune cell populations and their functional and molecular features, with the aim of studying immune mechanisms involved in lung cancer, sarcoidosis, and COPD, as well as factors associated with disease progression and treatment response. All medical care and treatment decisions remain independent of study participation.

SUMMARY:
This study aims to better understand the role of immune system cells in lung diseases such as lung cancer, sarcoidosis, and chronic obstructive pulmonary disease (COPD).

The investigators are studying how these immune cells can sometimes help the body defend itself, but in other cases may contribute to cancer growth or long-term lung inflammation.

Although recent treatments like immunotherapy have improved cancer care, only a small proportion of patients currently benefit from these therapies. One goal of this research is to understand why some patients do not respond or develop resistance to treatment.

The knowledge gained from this study may help researchers develop more effective and personalized treatments for people with lung diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung cancer
* Presence of precancerous lung lesions
* Patients with a chronic inflammatory lung disease (sarcoidosis or chronic obstructive pulmonary disease [COPD]) prior to any treatment
* Control group: individuals without known lung disease
* Children and adolescents weighing ≥ 10 kg with genetically confirmed chronic granulomatous disease (CGD)
* Adults scheduled to undergo orthopedic surgery during which a bone marrow sample will be collected

Exclusion Criteria:

* Systemic corticosteroid therapy > 10 mg/day prednisone (or equivalent)
* Acute infection at the time of inclusion
* Refusal or inability to provide informed consent (or assent, when applicable)
* Chronic inflammatory lung disease currently treated with immunosuppressive therapy

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 425 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2032-02-17 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Throughout the entire study, approximately during 7 years
  median Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Frank Aboubakar Nana, MD; PhD, Study Director — Cliniques universistaires saint Luc
Locations (1):
- Cliniques universitaires saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Desai A, Prasad V. Low-Dose Computed Tomographic Screening for Lung Cancer: Time to Implement or Unresolved Questions? J Gen Intern Med. 2021 Oct;36(10):3202-3204. doi: 10.1007/s11606-021-06806-5. Epub 2021 Apr 26. No abstract available. PMID 33904047
- [Result] Haslam A, Prasad V. Estimation of the Percentage of US Patients With Cancer Who Are Eligible for and Respond to Checkpoint Inhibitor Immunotherapy Drugs. JAMA Netw Open. 2019 May 3;2(5):e192535. doi: 10.1001/jamanetworkopen.2019.2535. PMID 31050774
- [Result] Delhez N, Aboubakar Nana F, Houbion C, Bayard A, Bruger A, Vanhaver C, Brandau S, van der Bruggen P, Hirsch T. Deciphering neutrophil heterogeneity in human blood and tumors: Methods for isolating neutrophils and assessing their effect on T-cell proliferation. Methods Cell Biol. 2025;191:151-196. doi: 10.1016/bs.mcb.2024.10.010. Epub 2024 Nov 25. PMID 39824555
- [Result] Bruger AM, Dorhoi A, Esendagli G, Barczyk-Kahlert K, van der Bruggen P, Lipoldova M, Perecko T, Santibanez J, Saraiva M, Van Ginderachter JA, Brandau S. How to measure the immunosuppressive activity of MDSC: assays, problems and potential solutions. Cancer Immunol Immunother. 2019 Apr;68(4):631-644. doi: 10.1007/s00262-018-2170-8. Epub 2018 May 21. PMID 29785656
- [Result] Vanhaver C, Aboubakar Nana F, Delhez N, Luyckx M, Hirsch T, Bayard A, Houbion C, Dauguet N, Brochier A, van der Bruggen P, Bruger AM. Immunosuppressive low-density neutrophils in the blood of cancer patients display a mature phenotype. Life Sci Alliance. 2023 Nov 6;7(1):e202302332. doi: 10.26508/lsa.202302332. Print 2024 Jan. PMID 37931958